CLINICAL TRIAL: NCT01711125
Title: Exploring the Efficacy and Biobehavioural Basis of Baclofen in the Treatment of Alcoholic Liver Disease
Brief Title: Baclofen in the Treatment of Alcohol Dependence With or Without Alcoholic Liver Disease
Acronym: BacALD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: South West Sydney Local Health District (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); University of Sydney (Other)
Responsible Party: Principal Investigator, Professor Paul Haber, Clinica Director, South West Sydney Local Health District
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X11-0154
Record Dates: First submitted 2012-10-16; First posted 2012-10-22 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Alcoholic Liver Disease; Alcohol Dependence
MeSH Terms: conditions — Liver Diseases, Alcoholic; Alcoholism | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): Baclofen low dose
  Interventions: Drug: Baclofen 30mg/day
- Arm 2 (Experimental): Baclofen high dose
  Interventions: Drug: Baclofen 75mg/day
- Arm 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen 30mg/day — 30mg/day 10 mg t.i.d
  Arms: Arm 1
Drug: Baclofen 75mg/day — 75mg/day 25 mg t.i.d
  Arms: Arm 2
Drug: Placebo — Placebo 3 matched tabs/day
  Arms: Arm 3

SUMMARY:
To explore the effectiveness and biobehavioural basis of baclofen in improving treatment outcomes for alcohol dependence in people with or without alcoholic cirrhosis in a double-blind randomised placebo-controlled trial.

DETAILED DESCRIPTION:
This is a double-blind randomised placebo-controlled study investigating the efficacy of baclofen for the treatment of alcohol dependence in patients with alcoholic liver disease. Medications will be given for 12 weeks, with a further 6 months follow-up. Both male and female participants will be recruited to this study. Trial patients will be randomised to one of three treatment groups: (1) baclofen 30mg/day (10 mg t.i.d), (2) baclofen 75mg/day (25 mg t.i.d) or (3) Placebo (3 matched tabs/day).

This study will also include a second, parallel group of patients with alcohol dependence (non alcoholic-liver disease patients) that will undergo the trial protocol as described above. These patients will be randomised according to a separate list into one of three treatment groups: (1) baclofen 30mg/day (10 mg t.i.d), (2) baclofen 75mg/day (25 mg t.i.d) or (3) Placebo (3 matched tabs/day).

ELIGIBILITY:
Inclusion Criteria:

* ALD (for trial group 1), defined as the presence of symptoms and/or signs referable to liver disease with or without cirrhosis, in which alcohol use is considered to play a major aetiological role. Alcohol use will have exceeded an average of 60g/day in women and 80g/day in men for >10 years.
* Alcohol dependence according to the ICD-10 criteria (for both trial 1 and 2)
* Adequate cognition and English language skills to give valid consent and complete research interviews
* Willingness to give written informed consent
* Abstinence from alcohol for between 3 and 21 days
* Resolution of any clinically evident alcohol withdrawal (CIWA-AR)

Exclusion Criteria:

* Active major psychological disorder associated with psychosis or significant suicide risk
* Pregnancy or lactation
* Concurrent use of any psychotropic medication other than antidepressants
* Substance use other than nicotine if unstable
* Clinical evidence of persisting hepatic encephalopathy
* Pending incarceration
* Lack of stable housing
* Active peptic ulcers
* Unstable diabetes mellitus

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
alcohol consumption | 12 weeks
  as measured by the number of days abstinent, number of heavy drinking days, time to relapse, time to lapse and number of drinks per drinking day

SECONDARY OUTCOMES:
clinical markers of liver injury | 12 weeks
incidence of hepatic side effects | 12 weeks
craving for alcohol | 12 weeks
early termination due to side effects | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Haber, MBBS, Principal Investigator — Sydney Local Health District; Andrew Baillie, PhD, Principal Investigator — Macquarie University; Kirsten C Morley, PhD, Principal Investigator — University of Sydney
Locations (1):
- Drug Health Services, Royal Prince Alfred Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Morley KC, Louie E, Hurzeler T, Baillie A, Dore G, Phung N, Haber PS. Sex as a Potential Moderator for Baclofen Response in the Treatment of Alcohol Dependence. Front Glob Womens Health. 2022 Mar 29;3:807269. doi: 10.3389/fgwh.2022.807269. eCollection 2022. PMID 35425938
- [Derived] Logge WB, Morris RW, Baillie AJ, Haber PS, Morley KC. Baclofen attenuates fMRI alcohol cue reactivity in treatment-seeking alcohol dependent individuals. Psychopharmacology (Berl). 2021 May;238(5):1291-1302. doi: 10.1007/s00213-019-05192-5. Epub 2019 Feb 20. PMID 30788529
- [Derived] Morley KC, Lagopoulos J, Logge W, Baillie A, Adams C, Haber PS. Brain GABA levels are reduced in alcoholic liver disease: A proton magnetic resonance spectroscopy study. Addict Biol. 2020 Jan;25(1):e12702. doi: 10.1111/adb.12702. Epub 2018 Dec 18. PMID 30561840
- [Derived] Heng S, Jamshidi N, Baillie A, Louie E, Dore G, Phung N, Haber PS, Morley KC. Baclofen Response in Alcohol Dependent Patients Concurrently Receiving Antidepressants: Secondary Analysis From the BacALD Study. Front Psychiatry. 2018 Nov 19;9:576. doi: 10.3389/fpsyt.2018.00576. eCollection 2018. PMID 30524317
- [Derived] Morley KC, Baillie A, Fraser I, Furneaux-Bate A, Dore G, Roberts M, Abdalla A, Phung N, Haber PS. Baclofen in the treatment of alcohol dependence with or without liver disease: multisite, randomised, double-blind, placebo-controlled trial. Br J Psychiatry. 2018 Jun;212(6):362-369. doi: 10.1192/bjp.2018.13. Epub 2018 May 2. PMID 29716670
- [Derived] Morley KC, Leung S, Baillie A, Haber PS. The efficacy and biobehavioural basis of baclofen in the treatment of alcoholic liver disease (BacALD): study protocol for a randomised controlled trial. Contemp Clin Trials. 2013 Nov;36(2):348-55. doi: 10.1016/j.cct.2013.08.002. Epub 2013 Aug 9. PMID 23939511